CLINICAL TRIAL: NCT06002373
Title: Reliability Of Artificial Intelligence for Treatment Decision Recommendation of Adult Skeletal Class III Patients: A Diagnostic Test Accuracy Study
Brief Title: Assessment of Artificial Intelligence for Treatment Decision Recommendation of Adult Skeletal Class III Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Abd El-Monem Nasr, Principal Investigator, Cairo University
Other Study IDs: 8114
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Skeletal Dysplasia; Reverse Overjet
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study titled "Reliability Of Artificial Intelligence for Treatment Decision Recommendation of Adult Skeletal Class III Patients" aims to assess the accuracy and dependability of artificial intelligence (AI) in providing treatment decision recommendations for adult patients with skeletal Class III malocclusion. Skeletal Class III malocclusion is characterized by an underdeveloped upper jaw or an overdeveloped lower jaw, leading to facial and dental irregularities. The study focuses on evaluating whether AI-based recommendations can reliably guide orthodontic treatment planning for this specific patient group.

This diagnostic test accuracy study involves collecting a diverse dataset of adult patients diagnosed with skeletal Class III malocclusion. AI algorithms will be trained on this dataset using various clinical and radiographic parameters to learn patterns and make treatment recommendations. The study will then compare the AI-generated treatment recommendations to those provided by experienced orthodontists.

Key aspects of the study include:

AI Reliability: The primary objective is to assess how consistently and accurately the AI system can recommend appropriate treatment decisions for adult skeletal Class III patients.

Diagnostic Test Accuracy: The study will determine the sensitivity, specificity, positive predictive value, and negative predictive value of the AI-generated treatment recommendations. This analysis will highlight the AI's ability to correctly identify patients who require specific treatment interventions.

Clinical Validity: Researchers will investigate whether the AI recommendations align with the decisions made by experienced orthodontists. This assessment is crucial to establish the AI system's clinical applicability.

Potential Benefits: If the AI system proves reliable and accurate, it could offer a time-efficient and standardized method for treatment decision support, aiding orthodontists in providing personalized care to adult skeletal Class III patients.

By conducting this study, researchers aim to contribute to the advancement of AI-assisted medical decision-making within the field of orthodontics. Successful outcomes would have the potential to revolutionize treatment planning processes, improve patient outcomes, and provide a valuable tool for orthodontists to make informed treatment decisions for adult skeletal Class III patients

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients with CVMI 6.
* Skeletal class III patients
* No congenital deformity, syndrome, or cleft.
* No previous surgical intervention
* No mandibular transverse functional shift.
* Normal overjet, overbite after completion of treatment.
* Patients with well finished occlusion.
* Patients who have achieved adequate functional and aesthetic results at the end of their treatment.
* Good quality initial and final lateral cephalometric radiographs.
* No sex predilection.

Exclusion Criteria:

* Adolescents and skeletally immature patients.
* Patients with pseudo class III.
* Syndromic patients.
* Patients with facial deformity at the naso-maxillary complex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with skeletal Class III malocclusion
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity | 1 month
  the difference in sensitivity and specificity between the treatment decisions taken by the clinicians in comparison to those provided by the artificial intelligence software

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt